CLINICAL TRIAL: NCT03459755
Title: Evaluating Race Specific AGE Accumulation As a Behavioral Biomarker That Can Reflect Optimal Health in Prostate Cancer Survivors
Brief Title: Evaluating Race Specific AGE Accumulation As a Behavioral Biomarker Prostate Cancer Survivors
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: investigator decision
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 102805; Pro00071004 (Other: Medical University of South Carolina)
Record Dates: First submitted 2018-02-27; First posted 2018-03-09 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lifestyle Intervention (Experimental): Patients assigned to the Physical Activity arm will undergo exercise testing protocol and have supervised physical activity interventions while on study. Patients will also complete questionnaires and have research blood drawn.
  Interventions: Behavioral: Physical Activity
- Usual care (No Intervention): Patients will complete questionnaires and have research blood drawn.

INTERVENTIONS:
Behavioral: Physical Activity — Patients will have a baseline assessment by undergoing a maximal exercise testing protocol.
  For 12 weeks, patients will participate in an exercise session 3 days per week
  The patient will then enter a 12 week "Step Down" program in which the number of sessions is decreased to every week, then every 3 weeks.
  After the second 12-week period, the patient will enter a 28-week follow up period of unsupervised exercise.
  Arms: Lifestyle Intervention

SUMMARY:
The purpose of this study is to show that reduction in advanced glycation end-products (AGEs) is associated with the beneficial regulation of receptor for AGE (RAGE) mediated tumor response which may correlate with improved quality of life in PCa survivors. AGEs are produced by the body and are affected by lifestyle, weight and diet.

ELIGIBILITY:
Inclusion Criteria:

1. Patient diagnosed with non-metastatic Stage I-III Prostate Cancer
2. Age 45 years and older
3. Within 12 months of first histologic prostate cancer diagnosis.
4. Completed planned chemotherapy and/or radiation therapy 4 weeks or more prior to study.
5. BMI > 25
6. ECOG Performance Status 0 or 1.
7. Access to a telephone.
8. Able to read and understand written and spoken English.
9. Participants must be accessible for treatment and follow-up and must sign informed consent.
10. Subjects with known diabetes are permitted. However, they must be under active treatment for this condition.
11. Participants must past the cardiac rehabilitation center stress test.

Exclusion Criteria:

1. Planned enrollment in other formalized physical activity or diet counseling program during the 12 weeks of study
2. Received chemotherapy or radiation therapy within 4 weeks of enrollment
3. Had previous weight loss surgery (e.g. gastric bypass, sleeve gastrectomy and biliary pancreatic diversion).
4. Previously participated in Cardiac-Rehab
5. Have constrained mobility secondary to problems with balance, bone and/or joint disease
6. Have unstable angina or cardiovascular disease that prohibits exercise.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11-27 (Actual); Primary Completion 2019-11-27 (Actual); Study Completion 2019-11-27 (Actual)

PRIMARY OUTCOMES:
Compare RAGE response (measured in the blood) to changes in Quality of Life using the EORTC QLQ-30 questionnaire. | From baseline to up to 52 weeks
Compare RAGE response (measured in the blood) to changes in Quality of Life using the CES-D questionnaire. | From baseline to up to 52 weeks

SECONDARY OUTCOMES:
Effect of Lifestyle intervention (physical activity and diet) on AGE levels measured in the blood | From baseline up to 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David Turner, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States